CLINICAL TRIAL: NCT04644575
Title: A Phase 3 Open-label, Multicenter Study of the Long-term Safety and Efficacy of Intravenous Recombinant Coagulation Factor VIII Fc-von Willebrand Factor-XTEN Fusion Protein (rFVIIIFc-VWF-XTEN; BIVV001) in Previously Treated Patients With Severe Hemophilia A
Brief Title: Long-term Safety and Efficacy of Efanesoctocog Alfa (BIVV001) in Previously Treated Patients With Hemophilia A
Acronym: XTEND-ed
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS16294; U1111-1244-0517 (Registry Identifier: ICTRP); 2023-508929-27-00 (Registry Identifier: CTIS); 2020-002215-22 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-11-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BIVV001

STUDY DESIGN:
Intervention Model Description: It is a 3-arm study with single intervention
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Previously treated in BIVV001 study (Experimental): This arm includes participants who have completed study EFC16293 or study EFC16295, participants who have completed Arm B or Arm C of this study (LTS16294) and roll over into Arm A, and participants who have completed any other potential BIVV001 study. Participants in this arm will continue receiving BIVV001 prophylaxis treatment once weekly (QW) for a total of 100 exposure days (EDs) cumulative from the parent study and this study. Participants will have the opportunity to continue in this study for up to 4 years, unless BIVV001 is commercially available in their applicable participating country.
  Interventions: Drug: efanesoctocog alfa (BIVV001)
- Arm B: Newly initiated (China Only) in BIVV001 (Experimental): This arm includes Chinese participants of any age who will be newly initiated on BIVV001 prophylaxis treatment once-weekly (QW) for 52 weeks. After 52 weeks of treatment in this arm B, participants will be able to roll over into arm A.
  Interventions: Drug: efanesoctocog alfa (BIVV001)
- Arm C: Newly initiated in BIVV001 with planned major surgery (Experimental): This arm includes participants of any age who will be newly initiated on BIVV001 prophylaxis treatment once-weekly (QW) and will undergo planned major surgery after at least 6 initial EDs with BIVV001, and within 26 weeks from Day 1. After 52 weeks of treatment in arm C, participants will be able to roll into arm A.
  Interventions: Drug: efanesoctocog alfa (BIVV001)

INTERVENTIONS:
Drug: efanesoctocog alfa (BIVV001) — Pharmaceutical form:Solution for Injection Route of administration: Intravenous

SUMMARY:
Primary Objective:

- To evaluate the long-term safety of BIVV001 in previously treated subjects with hemophilia A

Secondary Objectives:

* To evaluate the efficacy of BIVV001 as a prophylaxis treatment.
* To evaluate the efficacy of BIVV001 in the treatment of bleeding episodes.
* To evaluate BIVV001 consumption for prevention and treatment of bleeding episodes.
* To evaluate the effect of BIVV001 prophylaxis on joint health outcomes.
* To evaluate the effect of BIVV001 prophylaxis on Quality of Life (QoL) outcomes.
* To evaluate the safety and tolerability of BIVV001 treatment.
* To assess the PK of BIVV001 based on the one stage activated partial thromboplastin time (aPTT) and two-stage chromogenic FVIII activity assays (only applicable to Arm B).
* To evaluate the efficacy of BIVV001 for perioperative management

DETAILED DESCRIPTION:
Participants will receive BIVV001 once weekly for a total of at least 100 exposure days to BIVV001 (including exposure during a BIVV001 parent study, if applicable). Participants will have the opportunity to continue in this study for up to 4 years, unless BIVV001 is commercially available in their applicable participating country.

ELIGIBILITY:
Inclusion criteria :

* For participants rolling over into Arm A

  * Participants who have completed the studies EFC16923, EFC16925, Arm B or Arm C of the current study, or any other potential BIVV001 study.
  * Male or Female
* For participants new to BIVV001 (Arm B and C)

  * Participants who have severe hemophilia A, defined as <1 IU/dL (<1%) endogenous FVIII activity as documented either by central laboratory testing at screening or in historical medical records from a clinical laboratory demonstrating <1% FVIII coagulant activity (FVIII:C) or a documented genotype known to produce severe hemophilia A.
  * Previous treatment for hemophilia A (prophylaxis or on-demand) with any recombinant and/or plasma-derived FVIII, or cryoprecipitate for at least 150 EDs or 50 EDs for participants aged <6 years.
  * Platelet count ≥100 000 cells/μL at screening.
  * A participant known to be human immunodeficiency virus (HIV) antibody positive, either previously documented or identified from screening assessments, must have the following results prior to enrollment: CD4 lymphocyte count >200 cells/mm³ and viral load of <400 000 copies/mL
  * Male
  * Only for Arm B: Chinese participants
  * Only for Arm C: planned major surgery within 6 months after Day 1.

Exclusion criteria:

* For participants rolling over into Arm A

  * Positive inhibitor result, defined as ≥0.6 Bethesda units (BU)/mL.
  * Participation in another study.
* For participants new to BIVV001 (Arm B and Arm C)

  * Any concurrent clinically significant liver disease that, in the opinion of the Investigator, would make the participant unsuitable for enrollment. This may include, but is not limited to cirrhosis, portal hypertension, and acute hepatitis.
  * Serious active bacterial, fungal, or viral infection (other than chronic hepatitis or HIV) present within 30 days of screening.
  * Other known coagulation disorder(s) in addition to hemophilia A.
  * History of hypersensitivity or anaphylaxis associated with any FVIII product.
  * History of a positive inhibitor (to FVIII) test defined as ≥0.6 BU/mL, or any value greater than or equal to the lower sensitivity cut-off for laboratories with cut-offs for inhibitor detection between 0.7 and 1.0 BU/mL, or clinical signs or symptoms of decreased response to FVIII administrations. Family history of inhibitors will not exclude the participant.
  * Positive inhibitor test (FVIII) result, defined as ≥0.6 BU/mL at screening.
  * Treatment with acetylsalicylic acid (ASA) or antiplatelet agents that are not nonsteroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to screening.
  * Treatment with NSAIDs greater than the maximum dose specified in the regional prescribing information within 2 weeks prior to screening.
  * Systemic treatment within 12 weeks prior to Screening with chemotherapy and/or other immunosuppressive drugs (except for the treatment of hepatitis C virus [HCV] or HIV).
  * Emicizumab use within the 20 weeks prior to screening.
  * Major surgery within 8 weeks prior to screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the occurrence of inhibitor development (neutralizing antibodies detected against factor VIII [FVIII]) | Baseline to month 48
  The number of participants with the occurrence of inhibitor development (neuatralizing antibodies detected against factor VIII [FVIII]) as determined via the Nijmegen modified Bethesda assay.

SECONDARY OUTCOMES:
Annual bleeding rate (ABR) | Baseline to month 48
  Annualized bleeding rate (ABR) for treated bleeding episodes and all bleeding episodes (including untreated bleeds).
Annualized bleeding rate (ABR) by type of bleed | Baseline to month 48
  Annualized bleeding rate (ABR) by type during prophylaxis treatment per study arm and parent study.
Annualized bleeding rate (ABR) by location | Baseline to month 48
  Annualized bleeding rate (ABR) by location during prophylaxis treatment per study arm and parent study.
Percentage of patients who maintain factor VIII (FVIII) above prespecified activity levels | Baseline to month 48
  Percentage of participants who maintain factor VIII (FVIII) activity levels over 7 days post dose during prophylaxis treatment per study arm and per parent study or arm.
Number of injections and dose of BIVV0001 to treat a bleeding episode | Month 48
Percentage of bleeding episode treated with a single injection of BIVV001 | Month 48
Assessment of response to BIVV001 treatment of individual bleeding episodes | Baseline to month 48
  Assessment of response to BIVV001 treatment of individual bleeding episodes based on the International Society on Thrombosis and Haemostasis (ISTH) 4-point response scale
Physician's global assessment (PGA) of participants response to BIVV001 | Baseline to month 48
  Physician's global assessment (PGA) of participant's response to BIVV001 treatment based on a 4-point response scale .
Total annualized BIVV001 consumption | Baseline to month 48
  Total annualized BIVV001 consumption per participant during prophylaxis treatment
Annualized joint bleeding rate (AJBR) | Baseline to month 48
Target joint resolution | Month 48
  Target joint development, resolution and maintenance of target joint resolution based on ISTH criteria.
Change from baseline in Hemophilia Joint Health Score (HJHS) | Baseline to month 48
  Change from Baseline to the end of study visit in total score and domain scores (eg, swelling and strength) assessed by the Hemophilia Joint Health Score (HJHS)
Change from baseline in PROMIS-SF Physical Function | Baseline to month 48
  Change in Quality of Life (QoL) measures from baseline to end of study visit per study arm and per parent study arm: PROMIS-SF Physical Function (participants aged ≥18 years old).)
Change from baseline in Haem-A-QoL total score and physical health score | Baseline to month 48
  Change from baseline in Haemophilia QoL Questionnaire for Adults (Haem-A-QoL) total and physical health domain score on participants aged ≥17 years old.
Change from baselin in Haemo-QoL total score and physical health score | Baseline to month 48
  Change from baseline in Haemophilia QoL Questionnaire for Children (Haemo-QoL) total and physical health domain score on participants aged ≥4 to 16 years old and parent proxy for participants aged ≥4 to to <12 years old.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Baseline to month 48
  Participants with occurrences of treatment emergent adverse events (AEs) and serious adverse events (SAEs).
Number of participants with the occurrence of embolic and thrombotic events | Baseline to month 48
  Participants with the occurrence of embolic and thrombotic events.
PK parameter: Maximum activity (Cmax) | Baseline to week 52
PK parameter: Elimination half-life (t1/2) | Baseline to week 26
PK parameter: Total clearance (CL) | Baseline to week 26
PK parameter: Total clearance at steady state (CLss) | Baseline to week 26
PK parameter: Accumulation index (AI) | Baseline to week 26
PK parameter: Area under the activity time curve (AUC) | Baseline to week 26
PK parameter: Volume of distribution at steady state (Vss) | Baseline to week 26
PK parameter: Mean residence time (MRT) | Baseline to week 26
PK parameter: Incremental recovery (IR) | Baseline to week 52
PK parameter: Trough activity (Ctrough) | Baseline to week 52
PK parameter: Time above FVIII activity levels | Baseline to week 26
Investigators' or Surgeons' assessment of participant's hemostatic response to BIVV001 treatment | Baseline to month 48
  Investigators' or Surgeons' assessment of participant's hemostatic response to BIVV001 treatment on the ISTH 4 point response for surgical procedures scale.
Number of injections and dose to maintain hemostasis during perioperative period for major surgery | Baseline to month 48
Total BIVV001 consumption during perioperative period for major surgery | Baseline to month 48
Number and type of blood component transfusions used during perioperative period for major surgery | Baseline to month 48
Estimated blood loss during perioperative period for major surgery | Baseline to month 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (85):
- United States (16):
  - Orthopaedic Institute for Children Site Number : 8400003, Los Angeles, California
  - Children's Hospital Los Angeles Site Number : 8400009, Los Angeles, California
  - University of California San Diego Site Number : 8400007, San Diego, California
  - University of Florida Health Site Number : 8400008, Gainesville, Florida
  - Children's Healthcare of Atlanta Site Number : 8400016, Atlanta, Georgia
  - Rush University Medical Center Site Number : 8400010, Chicago, Illinois
  - Children's Hospital Of Iowa Site Number : 8400011, Iowa City, Iowa
  - University of Michigan Medical Center Site Number : 8400006, Ann Arbor, Michigan
  - Michigan State University School Of Med Site Number : 8400002, East Lansing, Michigan
  - Hemostasis and Thrombosis Center of Nevada Site Number : 8400001, Las Vegas, Nevada
  - New York Presbyterian Hospital/Weill Cornell Medical Center Site Number : 8400017, New York, New York
  - East Carolina University -2390 Hemby Ln Site Number : 8400015, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center Site Number : 8400012, Cincinnati, Ohio
  - Children's Research Institute Site Number : 8400013, Columbus, Ohio
  - Bloodworks Northwest Site Number : 8400005, Seattle, Washington
  - Children's Hospital of Wisconsin Site Number : 8400014, Milwaukee, Wisconsin
- Argentina (3):
  - Investigational Site Number : 0320001, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320002, Godoy Cruz, Mendoza Province
  - Investigational Site Number : 0320003, Buenos Aires
- Australia (4):
  - Investigational Site Number : 0360004, Camperdown, New South Wales
  - Investigational Site Number : 0360001, Westmead, New South Wales
  - Investigational Site Number : 0360002, South Brisbane, Queensland
  - Investigational Site Number : 0360003, Murdoch, Western Australia
- Investigational Site Number : 0560003, Woluwe-Saint-Lambert, Belgium
- Hemocentro Campinas - UNICAMP Site Number : 0760001, Campinas, São Paulo, Brazil
- Bulgaria (2):
  - Investigational Site Number : 1000171, Plovdiv
  - Investigational Site Number : 1000172, Sofia
- Canada (4):
  - Investigational Site Number : 1240005, Hamilton, Ontario
  - Investigational Site Number : 1240004, Hamilton, Ontario
  - Investigational Site Number : 1240002, Ottawa, Ontario
  - Investigational Site Number : 1240001, Toronto, Ontario
- China (10):
  - Investigational Site Number : 1560002, Beijing
  - Investigational Site Number : 1560006, Beijing
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560003, Hangzhou
  - Investigational Site Number : 1560004, Hangzhou
  - Investigational Site Number : 1560005, Jinan
  - Investigational Site Number : 1560009, Kunming
  - Investigational Site Number : 1560010, Kunming
  - Investigational Site Number : 1560013, Lanzhou
  - Investigational Site Number : 1560007, Suzhou
- France (5):
  - Investigational Site Number : 2500005, Brest
  - Investigational Site Number : 2500004, Bron
  - Investigational Site Number : 2500001, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500003, Lille
  - Investigational Site Number : 2500006, Marseille
- Germany (4):
  - Investigational Site Number : 2760304, Berlin
  - Investigational Site Number : 2760302, Bonn
  - Investigational Site Number : 2760001, Frankfurt am Main
  - Investigational Site Number : 2760002, München
- Investigational Site Number : 3000001, Athens, Greece
- Hungary (3):
  - Investigational Site Number : 3480002, Budapest
  - Investigational Site Number : 3480004, Debrecen
  - Investigational Site Number : 3480005, Pécs
- Investigational Site Number : 3720001, Dublin, Ireland
- Italy (3):
  - Investigational Site Number : 3800002, Napoli, Campania
  - Investigational Site Number : 3800001, Milan
  - Investigational Site Number : 3800003, Vicenza
- Japan (6):
  - Investigational Site Number : 3920425, Nagoya, Aichi-ken
  - Investigational Site Number : 3920423, Kitakyushu-shi, Fukuoka
  - Investigational Site Number : 3920426, Kawasaki-shi, Kanagawa
  - Investigational Site Number : 3920422, Kashihara-Shi, Niigata
  - Investigational Site Number : 3920421, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920424, Suginami-ku, Tokyo
- Netherlands (2):
  - Investigational Site Number : 5280002, Amsterdam
  - Investigational Site Number : 5280001, Utrecht
- South Korea (3):
  - Investigational Site Number : 4100603, Daegu, Daegu
  - Investigational Site Number : 4100601, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100600, Seoul, Seoul-teukbyeolsi
- Spain (2):
  - Investigational Site Number : 7240002, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240001, Madrid, Madrid, Comunidad de
- Investigational Site Number : 7520001, Malmo, Sweden
- Investigational Site Number : 7560001, Zurich, Switzerland
- Taiwan (5):
  - Investigational Site Number : 1580005, Changhua County
  - Investigational Site Number : 1580001, Taichung
  - Investigational Site Number : 1580003, Taichung
  - Investigational Site Number : 1580002, Taipei
  - Investigational Site Number : 1580004, Taipei
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920004, Antalya
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920003, Izmir
- United Kingdom (4):
  - Investigational Site Number : 8260005, London, London, City of
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260003, Birmingham
  - Investigational Site Number : 8260004, Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Quintilla JM, de la Gala C, Berrueco R, Claverol J, Figueres B, Bergos A, Rodriguez L, Mora A, DiBiaso V, Llanos C, Nafria B. High-Fidelity Clinical Simulation to Improve a Pediatric Clinical Trial Design: Lessons Learned and Conceptualization of the Return on Investment (ROI) and Return on Engagement (ROE) Analysis. Paediatr Drugs. 2025 Jan;27(1):73-84. doi: 10.1007/s40272-024-00660-8. Epub 2024 Nov 25. PMID 39585605